CLINICAL TRIAL: NCT04183413
Title: Strengthening Primary Healthcare Delivery for Diabetes and Hypertension in Eswatini: A Cluster-randomized Trial
Brief Title: Strengthening Primary Healthcare Delivery for Diabetes and Hypertension in Eswatini
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Collaborators: Amsterdam Institute for Global Health and Development (Other); Swiss Tropical & Public Health Institute (Other); Clinton Health Access Initiative, Eswatini (Unknown); University of Göttingen (Other); University of Eswatini (Unknown); SWABCHA, Eswatini (Unknown); Diabetes Swaziland (Unknown)
Responsible Party: Principal Investigator, Till Bärnighausen, Prof. Dr. Dr. Till Bärnighausen, University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: WHO-PEN@Scale
Record Dates: First submitted 2019-11-22; First posted 2019-12-03 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Diabetes Mellitus; Hypertension
Keywords: Diabetes Mellitus; Diabetes; Hypertension; WHO-PEN; Health service decentralization; Community Health Worker; Eswatini; Swaziland; Scale-up; Implementation research; Cost-effectiveness; Mixed methods; Comorbidity; Non-Communicable Disease; Cardiovascular disease risk factors
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Noncommunicable Diseases | interventions — Cytidine Diphosphate

STUDY DESIGN:
Intervention Model Description: This is a parallel three-arm cluster-randomized trial without a baseline assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard of Care (No Intervention): Health services for diabetes and hypertension are provided as was the standard of care prior to the healthcare reform after the emergency decentralization motivated by the COVID-19 outbreak. Healthcare for diabetes and hypertension for complicated cases is provided through physician-led teams at hospitals and health centers. Healthcare for diabetes and hypertension for uncomplicated cases is provided at primary care clinics through nurses.
- DSD (Experimental): Clients are invited to participate in one of three Differentiated Service Delivery models tailored to their needs.
  Interventions: Other: DSD
- CDP (Experimental): Health services for diabetes and hypertension are provided in the scope of outreach activities set up on a monthly basis in communities.
  Interventions: Other: CDP

INTERVENTIONS:
Other: DSD — This intervention consist of three Differentiated Service Delivery Models in which stable clients can be enrolled. The fast-track model gives preferential treatment to enrolled clients. Clients arrive at clinics, usually early in the morning, and can see the nurse as well as collect their medication without queuing. This model mainly targets the working population. The facility-based treatment clubs consist of bimonthly meetings where clients meet in groups of approximately 20 members. They receive health counselling, risk factor screening and medication prescription. This model mainly targets clients living close to the facility. The community advisory groups consist of groups of up to six clients. Groups are equipped with a point of care blood pressure and blood glucose measurement devices. They take turns in collecting the medication for the entire group and meet on a monthly basis. This model targets clients in hard-to-reach areas.
  Arms: DSD
Other: CDP — Community Distribution Points are set up on a monthly basis in communities linked to the clinic. Healthcare staff sets up a temporary point of contact where clients can obtain screening for diabetes and hypertension, health counselling, referral to primary or tertiary facilities, and medication.
  Arms: CDP

SUMMARY:
The WHO-PEN@Scale project is a three-arm cluster-randomized trial that is investigating the population-level effects of a healthcare reform in Eswatini, which aims to strengthen primary care for diabetes and hypertension. Prior to the reform, healthcare for diabetes and hypertension was mostly provided through physician-led teams in hospital outpatient departments. The healthcare reform aims to strengthen the provision of nurse-led care for diabetes and hypertension in primary healthcare facilities and community health worker-led care for these conditions in the facilities' catchment areas. The reform will broadly be guided by the World Health Organization's "Package of Essential Noncommunicable Disease Interventions for Primary Health Care in Low-Resource Settings" (WHO-PEN). The trial will take place at 84 clusters (a primary healthcare facility and its catchment area) across the country.

ELIGIBILITY:
Inclusion criteria for the outcome assessment (household survey):

* Residing in one of the selected households
* Age ≥40 years

Exclusion criteria for the outcome assessment (household survey):

* Pregnant
* Inability to provide written informed consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3500 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-12-05 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Glycemic control (continuous) among adults with diabetes | 12 months
  Mean glycated haemoglobin (HbA1c) among adults aged 40 years and older with diabetes
Systolic blood pressure among adults with hypertension | 12 months
  Mean systolic blood pressure among adults aged 40 years and older with hypertension

SECONDARY OUTCOMES:
HbA1c among adults with diabetes or prediabetes | 12 months
  Mean glycated haemoglobin (HbA1c) among adults aged 40 years and older with diabetes or prediabetes
Glycemic control (binary) among adults with diabetes | 12 months
  The proportion of adults aged 40 years and older with diabetes who have an HbA1c less than 7.0%
Glycemic control (binary) among adults with diabetes or prediabetes | 12 months
  The proportion of adults aged 40 years and older with diabetes or prediabetes who have an HbA1c less than 7.0%
Awareness of one's diabetes diagnosis | 12 months
  The proportion of adults aged 40 years and older with diabetes who report to have been diagnosed with diabetes prior to the household survey
Awareness of one's diabetes or prediabetes diagnosis | 12 months
  The proportion of adults aged 40 years and older with diabetes or prediabetes who report to have been diagnosed with diabetes or prediabetes prior to the household survey
Probability of being treated for diabetes among adults with diabetes | 12 months
  The proportion of adults aged 40 years and older with diabetes who report to be taking medication for their diabetes
Probability of having been tested for diabetes among adults with diabetes | 12 months
  The proportion of adults aged 40 years and older with diabetes who report to have ever been tested for diabetes
Probability of having been tested for diabetes among adults with diabetes or prediabetes | 12 months
  The proportion of adults aged 40 years and older with diabetes or prediabetes who report to have ever been tested for diabetes
Probability of smoking among adults with diabetes, prediabetes, or hypertension | 12 months
  The proportion of adults aged 40 years and older with diabetes, prediabetes, or hypertension who report to be a current smoker
Time spent doing moderate- or vigorous-intensity exercise among adults with diabetes, prediabetes, or hypertension | 12 months
  The mean number of minutes in a typical week spent doing moderate- or vigorous-intensity exercise among adults aged 40 years and older with diabetes
Systolic blood pressure among adults with diabetes | 12 months
  Mean systolic blood pressure among adults aged 40 years and older with diabetes
Systolic blood pressure among adults with diabetes or prediabetes | 12 months
  Mean systolic blood pressure among adults aged 40 years and older with diabetes or prediabetes
Diastolic blood pressure among adults with diabetes | 12 months
  Mean diastolic blood pressure among adults aged 40 years and older with diabetes
Diastolic blood pressure among adults with diabetes or prediabetes | 12 months
  Mean diastolic blood pressure among adults aged 40 years and older with diabetes or prediabetes
Hypertension control (binary) among adults with hypertension | 12 months
  The proportion of adults aged 40 years and older with hypertension who have a systolic blood pressure <140 mm Hg and a diastolic blood pressure <90 mm Hg
Diastolic blood pressure among adults with hypertension | 12 months
  Mean diastolic blood pressure among adults aged 40 years and older with hypertension
Awareness of one's hypertension diagnosis | 12 months
  The proportion of adults aged 40 years and older with hypertension who report to have been diagnosed with hypertension prior to the household survey
Probability of being treated for hypertension among adults with hypertension | 12 months
  The proportion of adults aged 40 years and older with hypertension who report to be taking blood-pressure-lowering medication
Probability of having been tested for hypertension among adults with hypertension | 12 months
  The proportion of adults aged 40 years and older with hypertension who report to have ever had their blood pressure measured
Frequency of drinking alcohol in the past 12 months among adults with diabetes, prediabetes, or hypertension | 12 months
  The proportion of adults aged 40 years and older with diabetes, prediabetes, or hypertension who report to having drunk daily, 5-6 days per week, 3-4 days per week, 1-2 days per week, 1-3 days per month, less than once a month, or never over the past 12 months.
21. Knowledge on diabetes and hypertension among adults with diabetes, prediabetes, or hypertension | 12 months
  The proportion of adults aged 40 years and older with diabetes, prediabetes, or hypertension who correctly responded to each individual question on diabetes and hypertension related knowledge.

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Geldsetzer, MD ScD MPH, Principal Investigator — Stanford University; Jan-Walter De Neve, MD ScD MPH, Principal Investigator — Heidelberg Institute of Global Health, Heidelberg University
Locations (1):
- Clinton Health Access Initiative, Mbabane, Eswatini

IPD SHARING:
Plan to Share IPD: Yes
No detailed IPD sharing plan has been developed yet.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code

REFERENCES:
- [Derived] Harkare HV, Osetinsky B, Ginindza N, Cindzi BT, Mncina N, Akomolafe B, Marowa LR, Ntshalintshali N, Tediosi F. Human and financial resource needs for universal access to WHO-PEN interventions for diabetes and hypertension care in Eswatini: results from a time-and-motion and bottom-up costing study. Hum Resour Health. 2024 May 27;22(1):32. doi: 10.1186/s12960-024-00913-0. PMID 38802811
- [Derived] Theilmann M, Ginindza N, Myeni J, Dlamini S, Cindzi BT, Dlamini D, Dlamini TL, Greve M, Harkare HV, Hleta M, Khumalo P, Kolbe LM, Lewin S, Marowa LR, Masuku S, Mavuso D, Molemans M, Ntshalintshali N, Nxumalo N, Osetinsky B, Pell C, Reis R, Shabalala F, Simelane BR, Stehr L, Tediosi F, van Leth F, De Neve JW, Barnighausen T, Geldsetzer P. Strengthening primary care for diabetes and hypertension in Eswatini: study protocol for a nationwide cluster-randomized controlled trial. Trials. 2023 Mar 22;24(1):210. doi: 10.1186/s13063-023-07096-4. PMID 36949485

DOCUMENTS (1):
  • Statistical Analysis Plan (2019-11-10): https://cdn.clinicaltrials.gov/large-docs/13/NCT04183413/SAP_000.pdf